CLINICAL TRIAL: NCT04964531
Title: Left Ventricular Remodeling After Transcatheter Closure of the Patent Ductus Arteriosus. Comparative Study Between Different Age Groups
Brief Title: Effect of PDA Closure on the Left Ventricular Remodeling
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ahmed Mohamed Moheb El-Din (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed Moheb El-Din, Assistant lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: speckle tracking, PDA
Record Dates: First submitted 2021-06-28; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Congenital Heart Defect; Patent Ductus Arteriosus
MeSH Terms: conditions — Heart Defects, Congenital; Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults: group of adults includes all patients aging 19 years or more
  Interventions: Other: speckle tracking echocardiography
- children: group of children includes all patients aging less than 19 years
  Interventions: Other: speckle tracking echocardiography

INTERVENTIONS:
Other: speckle tracking echocardiography — before and after closure of the PDA , echocardiographic loops of the apical 4, 3 , and 2 chamber will be acquired then processed by special software for measuring the speckle movements in the longitudinal and short axis views

SUMMARY:
failure of closure of the ductus arteriosus after birth results in a congenital anomaly known as patent ductus arteriosus. The large ductus can induce left side heart remodeling changes which could interfere with the normal cardiac function.

DETAILED DESCRIPTION:
Patent ductus arteriosus (PDA) is a congenital heart disease that represents 6-11% of all congenital heart diseases and is due to failure of spontaneous closure of a normal foetal duct called ductus arteriosus, that is a duct connecting the left pulmonary artery to the aorta, and it may result in LV volume overload , pulmonary overflow that may end with development of Eisenmenger syndrome. LV volume overload of the big ductus induce left heart remodeling changes in form of LA and LV dilatation, and LV hypertrophy to compensate for the increased wall stress. Some patients compensate well and remain asymptomatic, while others can't and develop manifestations of LV systolic dysfunction .

Traditional echocardiography is the main diagnostic tool for the PDA and assessment of its hemodynamic effect on the heart. speckle tracking echocardiography ( STE) is a relatively novel tool that can assess the LV function by tracking the speckles of the grey scale 2D images. Recent studies revealed good correlation between the LVEF measured by traditional echocardiography and global longitudinal strain (GLS) measured by STE , in addition to detection of subtle myocardial dysfunction by STE in patients with heart failure with preserved LVEF before frank LV systolic dysfunction is apparent clinically .

PDA closure should induce reverse remodelling with improvement of the left heart dimensions and function . Many studies in pediatrics showed deterioration of LVEF early after PDA closure followed by rapid recovery , while fewer studies showed late improvement of the LVEF in the adults .

ELIGIBILITY:
Inclusion Criteria:

* all patients who are candidate for transcatheter PDA closure.

Exclusion Criteria:

1. Patients with PDA dependent pulmonary circulation.
2. Patients with small sized PDA which is silent by auscultation.
3. Patients with large sized PDA which is unsuitable for Trans-catheter closure .
4. Patients with PDA and severe irreversible pulmonary hypertension (Eisenmenger's syndrome) (7).
5. Patients with active infection or active infective endarteritis.
6. Patients refusing the study.
7. Patients with DM, HTN and ischemic heart diseases.
8. Patients with associated congenital or acquired cardiac lesions that may interfere with LV mechanics.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: the study population will include all patients diagnosed as having patent ductus arteriosus and this ductus either hemodynamically insignificant but with audible murmur or this duct causes left heart volume overload symptoms
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
change of LV strain after transcatheter closure of the PDA | at base line, within 48 hours after closure of the duct then at three and six months
  Assess the change of left ventricular longitudinal and circumferential strain by speckle tracking echocardiography after PDA closure, and compare this change between the children and adults.

REFERENCES:
- [Background] Morton SU, Brodsky D. Fetal Physiology and the Transition to Extrauterine Life. Clin Perinatol. 2016 Sep;43(3):395-407. doi: 10.1016/j.clp.2016.04.001. Epub 2016 Jun 11. PMID 27524443
- [Background] Weir EK, Obreztchikova M, Vargese A, Cabrera JA, Peterson DA, Hong Z. Mechanisms of oxygen sensing: a key to therapy of pulmonary hypertension and patent ductus arteriosus. Br J Pharmacol. 2008 Oct;155(3):300-7. doi: 10.1038/bjp.2008.291. Epub 2008 Jul 21. PMID 18641675
- [Background] P S, Jose J, George OK. Contemporary outcomes of percutaneous closure of patent ductus arteriosus in adolescents and adults. Indian Heart J. 2018 Mar-Apr;70(2):308-315. doi: 10.1016/j.ihj.2017.08.001. Epub 2017 Aug 9. PMID 29716712
- [Background] Schneider DJ. The patent ductus arteriosus in term infants, children, and adults. Semin Perinatol. 2012 Apr;36(2):146-53. doi: 10.1053/j.semperi.2011.09.025. PMID 22414886
- [Background] Mor-Avi V, Lang RM, Badano LP, Belohlavek M, Cardim NM, Derumeaux G, Galderisi M, Marwick T, Nagueh SF, Sengupta PP, Sicari R, Smiseth OA, Smulevitz B, Takeuchi M, Thomas JD, Vannan M, Voigt JU, Zamorano JL. Current and evolving echocardiographic techniques for the quantitative evaluation of cardiac mechanics: ASE/EAE consensus statement on methodology and indications endorsed by the Japanese Society of Echocardiography. Eur J Echocardiogr. 2011 Mar;12(3):167-205. doi: 10.1093/ejechocard/jer021. PMID 21385887
- [Background] Mondillo S, Galderisi M, Mele D, Cameli M, Lomoriello VS, Zaca V, Ballo P, D'Andrea A, Muraru D, Losi M, Agricola E, D'Errico A, Buralli S, Sciomer S, Nistri S, Badano L; Echocardiography Study Group Of The Italian Society Of Cardiology (Rome, Italy). Speckle-tracking echocardiography: a new technique for assessing myocardial function. J Ultrasound Med. 2011 Jan;30(1):71-83. doi: 10.7863/jum.2011.30.1.71. PMID 21193707
- [Background] Edvardsen T, Helle-Valle T, Smiseth OA. Systolic dysfunction in heart failure with normal ejection fraction: speckle-tracking echocardiography. Prog Cardiovasc Dis. 2006 Nov-Dec;49(3):207-14. doi: 10.1016/j.pcad.2006.08.008. PMID 17084180
- [Background] Amoogzar H, Shakiba AM, Derakhshan D, Ajami G, Cheriki S, Borzouee M, Edraki MR, Mehdizadegan N. Evaluation of left ventricular function by tissue Doppler and speckle-derived strain rate echocardiography after percutaneous ductus closure. Pediatr Cardiol. 2015 Jan;36(1):219-25. doi: 10.1007/s00246-014-0989-0. Epub 2014 Aug 9. PMID 25107547
- [Background] Tilahun B, Tefera E. Transient left ventricular systolic dysfunction following surgical closure of large patent ductus arteriosus among children and adolescents operated at the cardiac centre, Ethiopia. J Cardiothorac Surg. 2013 May 31;8:139. doi: 10.1186/1749-8090-8-139. PMID 23721219
- [Background] Jeong YH, Yun TJ, Song JM, Park JJ, Seo DM, Koh JK, Lee SW, Kim MJ, Kang DH, Song JK. Left ventricular remodeling and change of systolic function after closure of patent ductus arteriosus in adults: device and surgical closure. Am Heart J. 2007 Sep;154(3):436-40. doi: 10.1016/j.ahj.2007.04.045. PMID 17719286
- [Background] Zhan Z, Guan L, Pan W, Zhang X, Zhang L, Zhou D, Ge J. Left ventricular size and function after percutaneous closure of patent ductus arteriosus in Chinese adults. Int J Cardiol. 2020 Sep 15;315:24-28. doi: 10.1016/j.ijcard.2020.04.060. Epub 2020 Apr 22. PMID 32333933
- [Background] Yasuhara J, Kuno T, Kumamoto T, Kojima T, Shimizu H, Yoshiba S, Kobayashi T, Sumitomo N. Comparison of transcatheter patent ductus arteriosus closure between children and adults. Heart Vessels. 2020 Nov;35(11):1605-1613. doi: 10.1007/s00380-020-01639-4. Epub 2020 Jun 3. PMID 32494943